CLINICAL TRIAL: NCT06667570
Title: Efficacy of the SALFOAM 3% Method Compared to the Conventional Polidocanol Foam Method (Tessari Method) for Treating Lower Limb Varicose Veins
Acronym: SALFOAM 3%
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lidiane Rocha (Other)
Responsible Party: Sponsor-Investigator, Lidiane Rocha, Principal Investigator, Science Valley Research Institute
Organization: Science Valley Research Institute (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SALFOAM 3%
Record Dates: First submitted 2024-10-28; First posted 2024-10-31 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Varicose Veins
Keywords: Chronic Venous Disease; Varicose Veins; Polidocanol Foam; Sclerotherapy; SALFOAM 3%; Tessari Method; Vein Occlusion; Hyperpigmentation
MeSH Terms: conditions — Varicose Veins; Hyperpigmentation | interventions — Control Groups

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SALFOAM 3% (Experimental): Participants in this group will receive a saline wash, followed by an injection of polidocanol 3% foam using the Tessari method, and extrinsic compression with Lidstop® over the treated vein. This is followed by the application of elastic compression stockings (20-30 mmHg) for 72 hours.
  Interventions: Procedure: SALFOAM 3%
- Tessari Method (Active Comparator): Participants in this group will receive the conventional Tessari method of polidocanol 3% foam injection, followed by compression with a dental roll and elastic compression stockings (20-30 mmHg) for 24 hours.
  Interventions: Procedure: Control Group

INTERVENTIONS:
Procedure: SALFOAM 3% — * Drug: Polidocanol 3%
  * Device: Lidstop®
  Arms: SALFOAM 3%
Procedure: Control Group — * Drug: Polidocanol 3%
  * Device: Standard compression with dental roll and elastic stockings
  Arms: Tessari Method

SUMMARY:
This clinical trial aims to assess the efficacy and safety of the SALFOAM 3% method, which involves saline wash, polidocanol 3% foam injection, and extrinsic compression using Lidstop®, in comparison with the conventional Tessari method for the treatment of lower limb varicose veins. The primary objective is to determine whether the SALFOAM 3% method results in better or equivalent vein occlusion rates and fewer adverse effects, such as hyperpigmentation, compared to the standard treatment.

DETAILED DESCRIPTION:
Chronic venous disease (CVD) is prevalent in approximately 38% of the adult population in Brazil, posing significant public health challenges due to its potential complications, including ulcerations and reduced quality of life. The SALFOAM 3% method is a novel approach that combines saline wash prior to polidocanol 3% foam sclerotherapy and extrinsic compression with Lidstop®, aiming to improve outcomes by reducing adverse effects such as hyperpigmentation and enhancing patient quality of life. This randomized controlled trial will compare the efficacy, safety, and quality of life outcomes of patients treated with the SALFOAM 3% method versus those treated with the conventional Tessari method for lower limb varicose veins.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 years or older with clinically confirmed varicose veins in the lower limbs by ultrasonography.
* All Fitzpatrick skin types (I-VI).
* Ability to provide written informed consent.

Exclusion Criteria:

* Pregnancy or breastfeeding.
* Known allergy or adverse reaction to polidocanol or similar agents.
* Active infection in the area of treatment.
* Immunosuppressed patients.
* Severe coagulopathies or a history of recent deep vein thrombosis or pulmonary embolism.
* Diagnosis of patent foramen ovale.
* CEAP classification VI (active venous ulcers).
* Use of medications that may interfere with the study outcomes.
* Inability to comply with the study protocol or refusal to participate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2024-10-25 (Actual); Primary Completion 2025-02-14 (Actual); Study Completion 2025-02-14 (Actual)

PRIMARY OUTCOMES:
Vein Occlusion Rate at 30 Days | 30 days post-procedure
  Vein occlusion will be measured using Doppler ultrasound to assess whether the treated veins are completely occluded, partially occluded, or not occluded at 30 days post-procedure.

SECONDARY OUTCOMES:
Hyperpigmentation Rate | 7 and 30 days post-procedure
  Incidence of hyperpigmentation will be evaluated using a 4-point scale (1 = absent, 2 = mild, 3 = moderate, 4 = severe) at 7 and 30 days post-procedure.

OTHER OUTCOMES:
Adverse Event Rate | 7 and 30 days post-procedure
  Incidence of adverse events, including thrombophlebitis, skin ulceration, and other complications, will be assessed through clinical and ultrasound evaluations.
Quality of Life Improvement | 30 days post-procedure
  Measured using the revised Venous Clinical Severity Score (rVCSS) to assess changes in the quality of life of participants at 30 days post-procedure. The total score ranges from a minimum of 0 to a maximum of 30 for a single limb. Minimum score: 0. This indicates the complete absence of symptoms or signs for all 10 characteristics. Maximum score: 30. This indicates the most severe symptoms and signs across all 10 characteristics.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital São Luiz Gonzaga, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No
De-identified individual participant data (IPD) will be shared after publication. Data sharing will include the study protocol, statistical analysis plan, and final dataset.

REFERENCES:
- [Background] Danneil O, Dorler M, Stockfleth E, Stucker M. Factors influencing superficial and deep vein thrombosis after foam sclerotherapy in varicose veins. J Dtsch Dermatol Ges. 2022 Jul;20(7):929-938. doi: 10.1111/ddg.14748. Epub 2022 Jun 12. PMID 35691945
- [Background] Rutherford RB, Padberg FT Jr, Comerota AJ, Kistner RL, Meissner MH, Moneta GL. Venous severity scoring: An adjunct to venous outcome assessment. J Vasc Surg. 2000 Jun;31(6):1307-12. doi: 10.1067/mva.2000.107094. PMID 10842165
- [Background] Wong M, Parsi K, Myers K, De Maeseneer M, Caprini J, Cavezzi A, Connor DE, Davies AH, Gianesini S, Gillet JL, Grondin L, Guex JJ, Hamel-Desnos C, Morrison N, Mosti G, Orrego A, Partsch H, Rabe E, Raymond-Martimbeau P, Schadeck M, Simkin R, Tessari L, Thibault PK, Ulloa JH, Whiteley M, Yamaki T, Zimmet S, Kang M, Vuong S, Yang A, Zhang L. Sclerotherapy of lower limb veins: Indications, contraindications and treatment strategies to prevent complications - A consensus document of the International Union of Phlebology-2023. Phlebology. 2023 May;38(4):205-258. doi: 10.1177/02683555231151350. Epub 2023 Mar 14. PMID 36916540
- [Background] Watson JJ, Mansour MA. Cosmetic sclerotherapy. J Vasc Surg Venous Lymphat Disord. 2017 May;5(3):437-445. doi: 10.1016/j.jvsv.2017.02.002. PMID 28411713
- [Background] Gloviczki P, Lawrence PF, Wasan SM, Meissner MH, Almeida J, Brown KR, Bush RL, Di Iorio M, Fish J, Fukaya E, Gloviczki ML, Hingorani A, Jayaraj A, Kolluri R, Murad MH, Obi AT, Ozsvath KJ, Singh MJ, Vayuvegula S, Welch HJ. The 2023 Society for Vascular Surgery, American Venous Forum, and American Vein and Lymphatic Society clinical practice guidelines for the management of varicose veins of the lower extremities. Part II: Endorsed by the Society of Interventional Radiology and the Society for Vascular Medicine. J Vasc Surg Venous Lymphat Disord. 2024 Jan;12(1):101670. doi: 10.1016/j.jvsv.2023.08.011. Epub 2023 Aug 29. PMID 37652254
- [Background] Vasquez MA, Rabe E, McLafferty RB, Shortell CK, Marston WA, Gillespie D, Meissner MH, Rutherford RB; American Venous Forum Ad Hoc Outcomes Working Group. Revision of the venous clinical severity score: venous outcomes consensus statement: special communication of the American Venous Forum Ad Hoc Outcomes Working Group. J Vasc Surg. 2010 Nov;52(5):1387-96. doi: 10.1016/j.jvs.2010.06.161. Epub 2010 Sep 27. PMID 20875713
- [Background] Hamel-Desnos CM, Guias BJ, Desnos PR, Mesgard A. Foam sclerotherapy of the saphenous veins: randomised controlled trial with or without compression. Eur J Vasc Endovasc Surg. 2010 Apr;39(4):500-7. doi: 10.1016/j.ejvs.2009.11.027. Epub 2010 Jan 25. PMID 20097585
- [Background] De Maeseneer MG, Kakkos SK, Aherne T, Baekgaard N, Black S, Blomgren L, Giannoukas A, Gohel M, de Graaf R, Hamel-Desnos C, Jawien A, Jaworucka-Kaczorowska A, Lattimer CR, Mosti G, Noppeney T, van Rijn MJ, Stansby G, Esvs Guidelines Committee, Kolh P, Bastos Goncalves F, Chakfe N, Coscas R, de Borst GJ, Dias NV, Hinchliffe RJ, Koncar IB, Lindholt JS, Trimarchi S, Tulamo R, Twine CP, Vermassen F, Wanhainen A, Document Reviewers, Bjorck M, Labropoulos N, Lurie F, Mansilha A, Nyamekye IK, Ramirez Ortega M, Ulloa JH, Urbanek T, van Rij AM, Vuylsteke ME. Editor's Choice - European Society for Vascular Surgery (ESVS) 2022 Clinical Practice Guidelines on the Management of Chronic Venous Disease of the Lower Limbs. Eur J Vasc Endovasc Surg. 2022 Feb;63(2):184-267. doi: 10.1016/j.ejvs.2021.12.024. Epub 2022 Jan 11. No abstract available. PMID 35027279